CLINICAL TRIAL: NCT00002615
Title: A RANDOMISED, CONTROLLED TRIAL OF PRE- AND POST-OPERATIVE CHEMOTHERAPY IN PATIENTS WITH OPERABLE GASTRIC CANCER
Brief Title: Surgery With or Without Combination Chemotherapy in Treating Patients With Stomach Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000063914; MRC-ST02; EU-94035
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-08

CONDITIONS: Gastric Cancer
Keywords: stage II gastric cancer; stage III gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Epirubicin; Fluorouracil

INTERVENTIONS:
Drug: cisplatin
Drug: epirubicin hydrochloride
Drug: fluorouracil
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not known whether receiving chemotherapy before surgery may be more effective than surgery alone in treating patients with stomach cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery plus combination chemotherapy with surgery alone in treating patients with stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival and quality of life of patients with resectable stage II or III adenocarcinoma of the stomach treated with epirubicin, cisplatin, and fluorouracil before and after resection vs resection alone.
* Determine the effect of perioperative chemotherapy on the resectability of gastric cancer in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center and performance status (0 vs 1).

* Arm I: Patients undergo radical total gastrectomy or radical subtotal distal gastrectomy, at the discretion of the surgeon, with perigastric lymph node dissection. Patients also may undergo lymphadenectomy at the discretion of the surgeon. At the beginning of the laparotomy, a pre-aortic, infra-colic node is sampled for staging purposes and frozen sections are examined during surgery. Patients who are found to have metastatic disease undergo palliative resection at the discretion of the surgeon and postoperative chemotherapy at the discretion of the oncologist.
* Arm II: Patients receive fluorouracil (5-FU) IV continuously for 3 weeks and cisplatin IV over 4 hours (beginning 4 hours after initiation of 5-FU infusion) and epirubicin IV on day 1 (ECF). Treatment continues every 3 weeks for 3 courses. Within 6 weeks after completion of course 3 and when blood counts recover, patients undergo resection as in arm I. Beginning within 4-6 weeks after surgery, patients receive 3 additional courses of ECF.

Quality of life is assessed at baseline, at completion of study therapy, and then every 6 months for 2 years.

Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven resectable stage II or III adenocarcinoma of the stomach
* No evidence of locally inoperable or distant metastases on chest x-ray and any combination of abdominal ultrasound, CT scan, or laparoscopy

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* WHO 0-1

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No clinical evidence of uncontrolled angina pectoris, cardiac failure, or significant uncontrolled cardiac arrhythmia

Other:

* No medical contraindication to study therapy
* No other prior malignancy except nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 1994-06; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H. Allum, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Epsom General Hospital, Epsom, Surrey, United Kingdom

REFERENCES:
- [Result] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Result] Cunningham D, Allum WH, Stenning SP, et al.: Perioperative chemotherapy in operable gastric and lower oesophageal cancer: final results of a randomised, controlled trial (the MAGIC trial, ISRCTN 93793971). [Abstract] J Clin Oncol 23 (Suppl 16): A-4001, 308s, 2005.
- [Result] Allum W, Cunningham D, Weeden S: Perioperative chemotherapy in operable gastric and lower oesophageal cancer: a randomised, controlled trial (the MAGIC trial, ISRCTN 93793971). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-998, 249, 2003.